CLINICAL TRIAL: NCT04583332
Title: Efficacy of Using Augmentative Alternative Communication for Functional Communication in Group Activities
Brief Title: Efficacy of AAC for Functional Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/00738 Sheeba Sharazi
Record Dates: First submitted 2020-10-06; First posted 2020-10-12 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Learning Disabilities; Cerebral Palsy; Down Syndrome
Keywords: AAC; Functional Communication; Group intervention
MeSH Terms: conditions — Learning Disabilities; Cerebral Palsy; Down Syndrome | interventions — Artifacts

STUDY DESIGN:
Intervention Model Description: Pre-post experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rhymes, Individual Items in Rhymes, Objects (Other): Existing method Post intervention
  Interventions: Other: Rhymes; Other: Individual Items in Rhymes; Other: Objects

INTERVENTIONS:
Other: Rhymes — Participants will be provided with a choice of 3 Nursery rhymes (Wheels on the bus, Old McDonald and Twinkle Twinkle Little Star) Objects pertaining to the 3 rhymes will be placed on a board Children will be given prompts as per their need and will be marked on the type of prompt given.
  These children will transit to pictures and Makaton symbols, if they are able to make choices using objects.
Other: Individual Items in Rhymes — Participants will be provided with a choice of 3 pictures within the initial choice making of the 2 Nursery rhymes (Wheels on the bus and Old McDonald ) Wheels on the Bus will include - mama/wipers/horn McDonalds - cow/dog/cat Objects pertaining to the 3 rhymes will be placed on a board Children will be given prompts as per their need and will be marked on the type of prompt given.
  These children will transit to pictures and Makaton symbols, if they are able to make choices using objects.
Other: Objects — Participants will be provided with 2,3 and 4 sensory objects. Participants will opt for an object by making a choice between these objects, if this is achieved then the child will be moved to picture level and symbol.

SUMMARY:
There is a considerable number children who are unable to speak, and our currently not being provided with any AAC options in their therapeutic facilities. The study aims to identify the current practice being employed with these children and then provide an AAC intervention for choice making with in group activities in the existing system, where the child is enrolled. Currently there is no indigenous evidence of AAC being employed effectively with these children. A pre- assessment will be carried out to establish the level of communication of the children. Intervention will be provided in a group for 6 weeks, three days a week, as these children already attend these groups.

DETAILED DESCRIPTION:
The study is a novel approach to intervention in Pakistan. There are currently no such studies conducted on intervention using AAC use in Pakistan. The objective of the the study are as follows

1. To compare establish current practices with AAC for choice making in group activities.
2. To determine the frequency of choice making in structured group activities.

Hypothesis:

Null Hypothesis:

The use of augmentative alternative communication does not increase functional communication in group activities.

Alternative Hypothesis:

The use of augmentative alternative communication increases functional communication in group activities.

Study Setting: Step to Learn School

Assessment: An assessment will be carried out using the online Communication Matrix to establish baseline communication skills of all the children. The children will also be assessed informally for their current means of communication in existing group activity at baseline, mid level (3 weeks) and at the end of the study (6 weeks).

Intervention: Intervention will (3 days a week for 6 weeks) be provided through objects, picture cards placed on a choice board. The choice will be given for Rhymes, Individual Rhymes & Sensory objects. Auditory, visual and tactile prompts will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Children with special needs
* Children not currently using any AAC

Exclusion Criteria:

* Children with any co-morbid conditions.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Self designed Questionnaire | 6 weeks
  Self designed questionnaire to address choice making in objects, pictures and symbols in three activities Rhymes, Items in Rhymes and Objects

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha K Butt, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Child Development Centre & Step to Learn School, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsahar Y, Hu S, Bouazza-Marouf K, Kerr D, Mansor A. Augmentative and Alternative Communication (AAC) Advances: A Review of Configurations for Individuals with a Speech Disability. Sensors (Basel). 2019 Apr 22;19(8):1911. doi: 10.3390/s19081911. PMID 31013673
- [Background] Meinzen-Derr J, Sheldon RM, Henry S, Grether SM, Smith LE, Mays L, Riddle I, Altaye M, Wiley S. Enhancing language in children who are deaf/hard-of-hearing using augmentative and alternative communication technology strategies. Int J Pediatr Otorhinolaryngol. 2019 Oct;125:23-31. doi: 10.1016/j.ijporl.2019.06.015. Epub 2019 Jun 20. PMID 31238158
- [Background] Nam S, Kim J, Sparks S. An Overview of Review Studies on Effectiveness of Major AAC Systems for Individuals with Developmental Disabilities Including Autism. Journal of Special Education Apprenticeship. 2018 Jun;7(2):n2.
- [Background] Schlosser RW, Wendt O. Effects of augmentative and alternative communication intervention on speech production in children with autism: a systematic review. Am J Speech Lang Pathol. 2008 Aug;17(3):212-30. doi: 10.1044/1058-0360(2008/021). PMID 18663107
- [Background] Lorah ER, Tincani M, Parnell A. Current trends in the use of handheld technology as a speech-generating device for children with autism. Behavior Analysis: Research and Practice. 2018 Aug;18(3):317.
- [Background] Waddington H, Sigafoos J, Lancioni GE, O'Reilly MF, van der Meer L, Carnett A, Stevens M, Roche L, Hodis F, Green VA, Sutherland D, Lang R, Marschik PB. Three children with autism spectrum disorder learn to perform a three-step communication sequence using an iPad(R)-based speech-generating device. Int J Dev Neurosci. 2014 Dec;39:59-67. doi: 10.1016/j.ijdevneu.2014.05.001. Epub 2014 May 10. PMID 24819024
- [Background] Roche L, Sigafoos J, Lancioni GE, O'Reilly MF, Schlosser RW, Stevens M, van der Meer L, Achmadi D, Kagohara D, James R, Carnett A, Hodis F, Green VA, Sutherland D, Lang R, Rispoli M, Machalicek W, Marschik PB. An evaluation of speech production in two boys with neurodevelopmental disorders who received communication intervention with a speech-generating device. Int J Dev Neurosci. 2014 Nov;38:10-6. doi: 10.1016/j.ijdevneu.2014.07.003. Epub 2014 Jul 21. PMID 25058915
- [Background] Stasolla F, De Pace C, Damiani R, Di Leone A, Albano V, Perilli V. Comparing PECS and VOCA to promote communication opportunities and to reduce stereotyped behaviors by three girls with Rett syndrome. Research in Autism Spectrum Disorders. 2014 Oct 1;8(10):1269-78.